CLINICAL TRIAL: NCT01012011
Title: Regulatory Post Marketing Surveillance Study on Nexavar®
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 14792; NX0910KR (Other: company internal)
Record Dates: First submitted 2009-11-10; First posted 2009-11-11 (Estimated); Last update posted 2015-09-21 (Estimated); Status verified 2015-09

CONDITIONS: Carcinoma, Hepatocellular; Carcinoma, Renal Cell
Keywords: Carcinoma, Hepatocellular; Carcinoma, Renal Cell
MeSH Terms: conditions — Carcinoma, Hepatocellular; Carcinoma, Renal Cell | interventions — Sorafenib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Sorafenib (Nexavar, BAY43-9006)

INTERVENTIONS:
Drug: Sorafenib (Nexavar, BAY43-9006) — Daily dose, dosage frequency and duration will be decided by physicians.

SUMMARY:
This surveillance are to identify problems/questions regarding adverse events, factors that are considered to affect on safety and efficacy in the clinical practice of using Nexavar

DETAILED DESCRIPTION:
The objectives of this surveillance are to identify problems/questions regarding the followings in the clinical practice of using Nexavar®.

1. Unknown adverse events (in particular, serious adverse events)
2. Identification of adverse events occurred in the real practice.
3. Factors that are considered to affect on safety.
4. Factors that are considered to affect on effectiveness

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of advanced RCC or HCC and decision taken by the physician to prescribe Nexavar.

Exclusion Criteria:

* Exclusion criteria must be read in conjunction with the local product information but patients who are participating in other interventional studies currently will be excluded.

Ages: 20 Years to 91 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosis of advanced renal cell carcinoma or hepatocellular carcinoma and decision taken by the physician to precribe Nexavar
Sampling Method: Non-Probability Sample
Enrollment: 2845 (Actual)
Dates: Start 2009-09; Primary Completion 2015-01 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Adverse events collection | From start of treatment to 4 weeks after discontinuation of treatment

SECONDARY OUTCOMES:
Duration of treatment, dosage and indication | Whole treatment period
Tumor status | Whole treatment period
Performance status | Whole treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, South Korea